CLINICAL TRIAL: NCT00914563
Title: An Optimizing of the Resuscitative Patterns by Use of Balanced Crystalloids and Colloids and the Non-Invasive Hemodynamic Monitoring
Brief Title: An Upgrading of the Resuscitative Patterns by Utilization of the Balanced Crystalloids and Synthetic Colloids and the Non-Invasive Hemodynamic Monitoring During Burn Shock
Acronym: FACT in BURNS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Faculty Hospital Kralovske Vinohrady, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FH Kralovske Vinohrady
Record Dates: First submitted 2009-05-28; First posted 2009-06-05 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Burns; Shock
Keywords: Burned shock; Volume resuscitative patterns; Non-invasive hemodynamic monitoring
MeSH Terms: conditions — Burns; Shock | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LIDCO (Experimental): The extensively burnt patients (age range 18-75 years) with second and the third degree burns, with TBSA above 15%, with or without inhalation injury will be included to the study. We will compare the standard monitored and volume resuscitated group of patients with the LIDCO monitored group. We will use in the LIDCO group the continuous real-time hemodynamic monitoring through transpulmonal lithium dilution additionally. The monitor Lithium Dilution Cardiac Output (LIDCO) Plus permits, through analysis of the arterial blood pressure trace, to acquire items about CO, SVR and DO2. In fluid resuscitation, we will use a combination of the balanced crystalloids and synthetic colloids (of the middle molecular weight) in the ratio 2 ml/kg/% TBSA: 1 ml/kg/% TBSA.
  Interventions: Device: LIDCO Lithium Dilution Cardiac Output
- Standard care (No Intervention): We will compare the standard monitored and volume resuscitated group of patients with the LIDCO monitored group. The control group will be composed of the patients supervised in a standard way, volume resuscitated according to the Brooke or Parkland formulas.
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: LIDCO Lithium Dilution Cardiac Output — Lithium Dilution Cardiac Output (LIDCO) Plus permits through analysis of the arterial blood pressure trace to acquire items about CO, SVR and DO2.
  Other Names: http://www.lidco-ir.co.uk/
  Arms: LIDCO
Other: Standard Care — We will compare the standard monitored and volume resuscitated group of patients with the LIDCO monitored group. The control group will be composed of the patients supervised in a standard way, volume resuscitated according to the Brooke or Parkland formulas.
  Other Names: Brooke or Parkland formulas
  Arms: Standard care

SUMMARY:
Fluid Therapy Lithium Dilution Cardiac Output (LIDCO) controlled trial in BURNS (FACT in BURNS) is a prospective randomized multicentric study.

Introduction: The goal of this trial is the verification, optional upgrading and optimizing of the resuscitative patterns in light of the new generation of balanced crystalloids and colloids and, by utilization the non-invasive hemodynamic monitoring LIDCO.

DETAILED DESCRIPTION:
Methods: The extensively burnt patients (age range 18-75 years) with second and the third degree burns, with TBSA above 15%, with or without inhalation injury will be included to the study within 2009-2010. The patients meeting inclusion criteria but with an adverse critical prognosis from the beginning of the hospitalization, with surgically insoluble extent of burns or the dialyzed patients will be excluded.The patients will be routinely monitored. We will use the continuous real-time hemodynamic monitoring through transpulmonal lithium dilution additionally. The monitor Lithium Dilution Cardiac Output (LIDCO) Plus permits through analysis of the arterial blood pressure trace to acquire items about CO, SVR and DO2 . In fluid resuscitation, we will use a combination of the balanced crystalloids and synthetic colloids (of the middle molecular weight) in the ratio 2 ml/kg/% TBSA : 1 ml/kg/% TBSA. The control group will be composed of the patients supervised in a standard way, volume resuscitated according to the Brooke or Parkland formulas. MAP > 65 torr, urine output 0,5 ml/kg/h, CI 2,5 - 4,0 l/min/m2, DO2I 500 - 600 ml/min/m2 are the goals.We will measure the levels of proANP (pro Natriuretic peptide) and Angiotensin Converting Enzyme (ACE) at artificial ventilated patients. The plasma ACE and proANP concentrations were measured by commercially available ELISA immunoassays.

Conclusions: We will evaluate the total fluid balance at day 1, 2 and cumulative fluid balance at day 7, reversal of organ dysfunction according to SOFA score at day 3 and 7 in both group. The days of invasive ventilatory support, length of ICU stay, ICU survival, total length of hospital stay and hospital survival are the additional endpoints.

ELIGIBILITY:
Inclusion Criteria:

* extensively burnt patients (age range 18-75 years) with second and third degree burns
* with TBSA above 15%
* with or without inhalation injury

Exclusion Criteria:

* patients meeting inclusion criteria but with an adverse critical prognosis from the beginning of hospitalization
* with surgically insoluble extent of burns
* dialyzed patients will be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The total fluid balance at day 1, 2 and cumulative fluid balance at day 7, reversal of organ dysfunction according to SOFA score at day 3 and 7 in both groups. | 2009-2010

SECONDARY OUTCOMES:
The days of invasive ventilatory support, length of ICU stay, ICU survival, total length of hospital stay and hospital survival. | 2009-2010

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Czechia

REFERENCES:
- [Background] Cartotto RC, Innes M, Musgrave MA, Gomez M, Cooper AB. How well does the Parkland formula estimate actual fluid resuscitation volumes? J Burn Care Rehabil. 2002 Jul-Aug;23(4):258-65. doi: 10.1097/00004630-200207000-00006. PMID 12142578
- [Background] Holm C, Melcer B, Horbrand F, von Donnersmarck GH, Muhlbauer W. The relationship between oxygen delivery and oxygen consumption during fluid resuscitation of burn-related shock. J Burn Care Rehabil. 2000 Mar-Apr;21(2):147-54. doi: 10.1097/00004630-200021020-00011. PMID 10752748
- [Background] Holm C, Melcer B, Horbrand F, Worl H, von Donnersmarck GH, Muhlbauer W. Intrathoracic blood volume as an end point in resuscitation of the severely burned: an observational study of 24 patients. J Trauma. 2000 Apr;48(4):728-34. doi: 10.1097/00005373-200004000-00023. PMID 10780609
- [Background] Holm C, Mayr M, Tegeler J, Horbrand F, Henckel von Donnersmarck G, Muhlbauer W, Pfeiffer UJ. A clinical randomized study on the effects of invasive monitoring on burn shock resuscitation. Burns. 2004 Dec;30(8):798-807. doi: 10.1016/j.burns.2004.06.016. PMID 15555792
- [Background] Huang Y, Yan B, Yang Z. Clinical study of a formula for delayed rapid fluid resuscitation for patients with burn shock. Burns. 2005 Aug;31(5):617-22. doi: 10.1016/j.burns.2005.02.002. PMID 15953681
- [Background] Ahrns KS. Trends in burn resuscitation: shifting the focus from fluids to adequate endpoint monitoring, edema control, and adjuvant therapies. Crit Care Nurs Clin North Am. 2004 Mar;16(1):75-98. doi: 10.1016/j.ccell.2003.09.007. PMID 15062415
- [Result] Mitra B, Fitzgerald M, Cameron P, Cleland H. Fluid resuscitation in major burns. ANZ J Surg. 2006 Jan-Feb;76(1-2):35-8. doi: 10.1111/j.1445-2197.2006.03641.x. PMID 16483293
- [Result] Berger MM, Bernath MA, Chiolero RL. Resuscitation, anaesthesia and analgesia of the burned patient. Curr Opin Anaesthesiol. 2001 Aug;14(4):431-5. doi: 10.1097/00001503-200108000-00009. PMID 17019126
- [Result] Czermak C, Hartmann B, Scheele S, Germann G, Kuntscher MV. [Burn shock fluid resuscitation and hemodynamic monitoring]. Chirurg. 2004 Jun;75(6):599-604. doi: 10.1007/s00104-004-0859-z. German. PMID 15103422